CLINICAL TRIAL: NCT06377943
Title: The Interaction Between Resting Metabolic Rate, Physical Activity and Thyroid Hormone in Females
Status: Completed | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, chief researcher, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-240415-H0718
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Thyroid; Physical Activities; Resting Energy Expenditure
MeSH Terms: conditions — Thyroid Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples and Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This Study is focused on the interaction between resting metabolic rate (RMR), physical activity (PA), and thyroid hormones (TH). TH controls almost all the cell activities of the body so, it is known as one of the major regulatory hormones. This is the reason for individuals who suffer from thyroid disorders show abnormal metabolism. Recently it was suggested that interindividual variations in thyroid hormone levels also influence daily physical activity.

DETAILED DESCRIPTION:
In this study, investigators will recruit adult females with a BMI ≥18.5. After the screening process, eligible volunteers will undergo certain measurements including body composition, resting metabolism daily physical activity, thyroid hormone levels, and total energy expenditure. The investigators will access the changes in resting metabolism and daily physical activities with the differences in thyroid hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥18;
* BMI≥18.5

Exclusion Criteria:

* Intended weight change exceeding 2kg within the past three months;
* Having any special medical diets or having eating disorders;
* Pregnant women or breastfeeding women;
* People who have metal implants in their bodies;
* Patients with metabolic diseases, infectious diseases, and genetic disorders such as hypothyroidism, and hyperthyroidism;
* Patients with a personal or family history of medullary thyroid carcinoma (MTC), or patients with rare type 2 multiple endocrine tumor syndrome (MEN2); People with a fear of needles (Trypanophobia), claustrophobia; People who are fear of blood (Hemophobia) or pathological hypotension;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study participants are adult healthy females.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-06-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Body weight | Measurements will take at the first day of the visit
  Subjects will be asked to fast overnight and weight will be measured using a calibrated Seca body weight scale first thing in the morning on subjects wearing light clothes and no shoes.
Height | Measurements will take at the first day of the visit
  Measured by seca 217 stable stadiometer. Subjects wearing no shoes.
Waist and Hip circumferences | Measurements will take at the first day of the visit
  Waist and Hip circumferences will be measured using a whole body laser scanner.
Fat mass | Measurements will take at the first day of the visit
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ) or DXA (Hologic).
Far free mass | Measurements will take at the first day of the visit
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980) or DXA (Hologic).
Bone mass | Measurements will take at the first day of the visit
  Bone mass will be measured by DXA (Hologic).
Resting Metabolism | Measurements will take at the first day of the visit.
  Resting energy expenditure will be measured using indirect calorimetry via a respiratory hood system (Cosmed). The subject attends the lab after an overnight fast. The person lies down on a flatbed and the hood is placed over their head. Metabolic rates (oxygen consumption and CO2 production) are monitored for 30 minutes. Calorimeters will be assessed with a turbine test to ensure the accuracy of measurements. Validation via an alcohol burn will be performed monthly.
Physical activity | Measurements last for 14 days
  Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 14 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day where the wear time is less than 10 hours. For a valid measure, the goal is to get at least 2 weekday and 2 weekend days.
Thyroid hormone | Blood samples will collect at the first day of the visit.
  Nurses will collect the blood samples on day 1. Levels of circulating thyroid hormones will be measured using radio immunoassay.
Resting Metabolism | measurements will take at the first day of visit
  The whole room calorimeter/metabolic chamber (OMNICAL, Maastricht instrument) will be used to measure resting metabolic rate. The metabolic chamber is a sealed room with a continuous gas supply (CO2- 0.80×10-2, O2 -18.00×10-2), providing subjects with 24-hour energy expenditure data. The total energy expenditure of the subjects in MJ/day was plotted against time in 30-minute intervals over 24 hours. The lowest and most stable energy expenditure during sleep time was considered the RMR of the subjects, which occurred from 2:00 am to 5:00 am.

SECONDARY OUTCOMES:
Total energy expenditure | Measurements take for 14 days
  Total energy expenditure (TEE) will be measured using the DLW method. Urine samples from all participants in the DLW subset will be stored at -20 oC and analyzed in the laboratory of Dr. John Speakman at the Shenzhen Institute of Advanced Technology, Chinese Academy of sciences. Isotopes will be measured in a benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation (Speakman et al 2021: Cell reports medicine). TEE will then be calculated using mean CO2 production using the Weir equation.
Total energy expenditure | Measurements take at the first day of the visit
  Total energy expenditure will be measured using the whole room calorimeter / metabolic chamber (OMNICAL, Maastricht instrument). The metabolic chamber is a sealed room with a continuous gas supply (CO2- 0.80×10-2, O2 -18.00×10-2), providing subjects with 24-hour energy expenditure data. The total energy expenditure was calculated by averaging the chamber's gaseous exchange using a 24-hour time window between 11.30 am and the next day around 3.00 pm.

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Study Chair — Shenzhen Institute of Advanced Technology, CAS
Locations (1):
- Shenzhen Institutes of Advanced Technology, Chinese Academy of Sciences, Shenzhen, Guangdong, China